CLINICAL TRIAL: NCT02858544
Title: Concussion in Motor Vehicle Accidents: The Concussion Identification Index
Acronym: CIDI
Status: Completed | Type: Observational
Sponsor: Clionsky Neuro Systems Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C-MVA
Record Dates: First submitted 2016-08-02; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Motor Vehicle Accidents; TBI (Traumatic Brain Injury); Brain Contusion; Brain Injuries; Cortical Contusion; Concussion Mild; Cerebral Concussion; Brain Concussion; Accidents, Traffic; Traffic Accidents; Traumatic Brain Injury With Brief Loss of Consciousness; Traumatic Brain Injury With no Loss of Consciousness; Traumatic Brain Injury With Loss of Consciousness
Keywords: Mild traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Contusion; Brain Injuries; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group1 - Validation Group: n=890 patients seen and evaluated for possible concussion after a motor vehicle accident. Patients with qualifying scores on the Concussion Identification Index will also complete the ImPACT.
  Interventions: Other: The Concussion Identification Index; Other: ImPACT
- Group 2 - Cross Validation Group: n=900 patients seen and evaluated for possible concussion after a motor vehicle accident. Patients with qualifying scores on the Concussion Identification Index will also complete the ImPACT.
  Interventions: Other: The Concussion Identification Index; Other: ImPACT

INTERVENTIONS:
Other: The Concussion Identification Index — Patient completion of the Concussion Identification Index, a report of crash characteristics, injuries sustained, and post-accident neurological signs and symptoms
Other: ImPACT — Patient- completed computerized neurocognitive test battery

SUMMARY:
The primary goal of this study is to provide clinicians with a brief, patient self-administer instrument yielding a single composite score that reliably correlates with objective findings on standardized neurocognitive assessment for concussion.

DETAILED DESCRIPTION:
This Phase 2 study, Concussion in Motor Vehicle Accidents - The Concussion Identification Index (CIDI), focuses on the psychometric properties of the relationship between acute injury events, i.e. head impact, loss of consciousness (LOC), and post-traumatic amnesia (PTA), commonly reported post-crash signs and symptoms, and neurocognitive outcomes.

Cohort 1 is the validation group and will be used to confirm the optimal cut-off score of the Concussion Identification Index (CIDI) with the score on the ImPACT.

Cohort 2 is the cross-validation group.

ELIGIBILITY:
Inclusion Criteria:

* Patients injured in a motor-vehicle related accident

Exclusion Criteria:

* Age younger than 10 years old or older than 60 years of age
* Patients who presented for initial evaluation of injuries greater than 90 days after MVA occurred
* Patients who declined to take a computerized neurocognitive test battery
* Patients who were not fluent in either English or Spanish

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cohort 1 - Validation Group: Consecutive patients who presented for care between November 1, 2013 and December 31, 2014 at the MVA Center for Rehabilitation, a public health clinic in Springfield, MA which provides specialized outpatient auto accident treatment and rehabilitation
  Cohort 2 - Cross Validation Group: Consecutive patients who presented for care between January 1, 2015 and June 30, 2016 at the MVA Center for Rehabilitation, a public health clinic in Springfield, MA
Sampling Method: Probability Sample
Enrollment: 1790 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Correlation - Concussion Identification Index score with ImPACT test score | Within 90 days of the accident

SECONDARY OUTCOMES:
Patient-completed one page questionnaire | Within 90 days of the accident
  The questionnaire is divided into two parts:
  The Injury Characteristics section: asks for a yes-no indication of whether 5 concussion-associated events/injuries occurred: striking the head, whiplash, loss of consciousness, being dazed, or having post-traumatic amnesia; and, whether or not the patient had already been given a diagnosis of concussion.
  The Concussive Symptoms section asks the patient to rate on a scale of 0-3 the presence and severity of 10 cognitive and emotional symptoms associated with a post-concussion diagnosis.
  The total numeric value for each patient is reported as an indexed score.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell I Clionsky, Ph.D, Principal Investigator — Clionsky Neuro Systems Inc.
Locations (1):
- Clionsky Neuro Systems, Inc., Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No